CLINICAL TRIAL: NCT03884400
Title: iSpecimen Network Distribution of Biospecimens From Biorepositories/Biobanks for Research Use
Brief Title: Distribution of Biospecimens From Biorepositories/Biobanks for Research Use
Status: Withdrawn | Type: Observational
Why Stopped: We have changed our research focus
Sponsor: iSpecimen Inc (Industry)
Responsible Party: Sponsor
Other Study IDs: ISPC-180828-DISTRIBUTION
Record Dates: First submitted 2019-03-18; First posted 2019-03-21 (Actual); Last update posted 2022-11-14 (Actual); Status verified 2022-11

CONDITIONS: Cancer; Pregnancy Related; Gastro-Intestinal Disorder; Cardio-Respiratory Distress; Women's Health: Endometriosis; Autoimmune Diseases; Nephritis; Healthy; Neuro-Degenerative Disease
Keywords: Observational
MeSH Terms: conditions — Neoplasms; Digestive System Diseases; Autoimmune Diseases; Nephritis | interventions — Phlebotomy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Subjects who have provided consent for specimen collection: Re-consent will not be required. This protocol allows distribution of the specimens following the terms agreed to by the subject in the original consent.
  Interventions: Procedure: Specimens obtained from surgical, phlebotomy or other non-invasive procedure

INTERVENTIONS:
Procedure: Specimens obtained from surgical, phlebotomy or other non-invasive procedure — Biospecimen Collection

SUMMARY:
This protocol seeks to assist biorepositories/biobanks in distributing their stored specimens and data to researchers that will actually utilize them to advance medicine and technology.

DETAILED DESCRIPTION:
iSpecimen has built a partner network comprised of supplying institutions that have ethically acquired human biospecimens and created biorepositories/biobanks to store the specimens and data.

Many of these biorepositories have protocols allowing for the collection of their samples but require an additional IRB or ethics review for the distribution of their samples.

This protocol establishes a method of such supply sites to allow their specimens to be distributed and used for research via iSpecimen's technology and network of research clients.

ELIGIBILITY:
Inclusion Criteria:

* Specimens and/or data from Biorepositories that have enrolled subjects that have provided consent for the specimens and de-identified data to be collected, stored and distributed.
* Specimens from biobanks that have collected materials and de-identified data under a waiver of consent
* Specimens from a biobank that meet the criteria for non human subject research under the common rule.

Exclusion Criteria:

* Specimens and/or that have been obtained from subjects without informed consent, nor waiver of consent or that do not meet the criteria for non human subject research under the common rule.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Diverse group of biorepositories with focus on cancer, neurodegenerative, pediatric, women's health and other cohorts.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Distribution of Biospecimens From Biorepositories/Biobanks for Research Use | 15 years
  The number of specimens and subjects distributed per disease will be measured and reported.

CONTACTS AND LOCATIONS:
Locations (1):
- iSpecimen, Lexington, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Website for specimen distribution — https://marketplace.ispecimen.com